CLINICAL TRIAL: NCT01419990
Title: Double-blind Placebo Controlled Dose-ranging Study for the Assessment of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Oral Dosing of GLPG0634 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Oral Doses of GLPG0634 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG0634-CL-102
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLPG0634 capsules (Experimental)
  Interventions: Drug: GLPG0634
- Placebo capsules (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG0634 — GLPG0634 300 mg oral capsules, qd, 10 days
  Arms: GLPG0634 capsules
Drug: GLPG0634 — GLPG0634 450 mg oral capsules, qd, 10 days
  Arms: GLPG0634 capsules
Drug: Placebo — Placebo oral capsules, qd, 10 days
  Arms: Placebo capsules

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of multiple ascending oral doses of GLPG0634 given to healthy subjects for 10 days compared to placebo.

During the course of the study, the amount of GLPG0634 present in the blood (pharmacokinetics) as well as the effects of GLPG0634 on mechanism of action-related parameters in the blood (pharmacodynamics) will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male, age 40-60 years
* BMI between 18-30 kg/m2

Exclusion Criteria:

* Any condition that might interfere with the procedures or tests in this study
* Drug or alcohol abuse
* Smoking

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | From screening up to 10 days after the last dose
  To evaluate the safety and tolerability of GLPG0634 in comparison with placebo after multiple oral doses in healthy subjects in terms of adverse events, physical examinations, vital signs, ECG and lab assessments

SECONDARY OUTCOMES:
Pharmacokinetics (PK) and pharmacodynamics (PD) | From first dose up to 10 days after the last dose
  To determine the plasma levels of GLPG0634 as a measure of PK and the levels of immune- and inflammation-related parameters as a measure of PD

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Vanhoutte, MD, Study Director — Galapagos NV; Lien Gheyle, MD, Principal Investigator — SGS Stuivenberg
Locations (1):
- SGS Stuivenberg, Antwerp, Antwerp, Belgium

REFERENCES:
- [Derived] Namour F, Diderichsen PM, Cox E, Vayssiere B, Van der Aa A, Tasset C, Van't Klooster G. Pharmacokinetics and Pharmacokinetic/Pharmacodynamic Modeling of Filgotinib (GLPG0634), a Selective JAK1 Inhibitor, in Support of Phase IIB Dose Selection. Clin Pharmacokinet. 2015 Aug;54(8):859-74. doi: 10.1007/s40262-015-0240-z. PMID 25681059